CLINICAL TRIAL: NCT02992678
Title: Prophylactic Treatment Pentoxifylline for the Prevention of Post-ERCP Pancreatitis
Brief Title: Pentoxifylline for the Prevention of PEP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: pentoxifylline-001
Record Dates: First submitted 2016-12-13; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline, 400 mg, 3 times daily by mouth the day before ERCP procedure. Subjects received up to a maximum of 3 doses.
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo, 400 mg, 3 times daily by mouth by mouth the day before ERCP procedure. . Subjects received up to a maximum of 3 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline, 400 mg, 3 times daily by mouth the day before ERCP procedure. Subjects received up to a maximum of 3 doses.
  Arms: Pentoxifylline
Drug: Placebo — Placebo, 400 mg, 3 times daily by mouth by mouth the day before ERCP procedure. . Subjects received up to a maximum of 3 doses.
  Arms: Placebo

SUMMARY:
Between December 2016 and June 2017, 110 consecutive patients older than 18 years who are scheduled to undergo diagnostic or therapeutic ERCP at the Anhui Provincial Hospital will be recruited for the study. Patients were randomized using opaque, sealed envelopes containing random numbers assigning them to treat with pentoxifylline (pentoxifylline group) or Placebo (placebo group) for preventing ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age > 18 years.
2. Normal amylase level before undergoing ERCP.
3. Signed inform consent form and agreed to follow-up on time.

Exclusion Criteria:

1. Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent.
2. Patients involved in other study within 60 days.
3. Billroth II or Roux-en-Y anatomy
4. Acute pancreatitis.
5. a history of previous ERCP
6. Pregnancy or history of allergy to pentoxifylline
7. Patient treated for arterial hypertension
8. Patient with severe coagulopathy
9. Patient with hyper sensibility of pentoxifylline
10. Nursing mothers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Acute Pancreatitis | 24 hours
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours, patients also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP (post-ERCP pancreatitis).

SECONDARY OUTCOMES:
The prophylaxis effect of pentoxifylline on post-ERCP pancreatitis in higher risk patients | 24 hours
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours in high risk patients, who also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis).

CONTACTS AND LOCATIONS:
Overall Officials: Shao Feng, MD, Principal Investigator — Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University
Locations (1):
- Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No